CLINICAL TRIAL: NCT06113718
Title: The Impact of Preoperative Bowel Exercise on Postoperative Bowel Functions in Gynecologic Malignancies
Acronym: IPBEPOBF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Celal Akdemir, Gynecologic Oncology Fellow, Tepecik Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TTRH
Record Dates: First submitted 2023-10-17; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Paralytic Ileus; Nausea; Defecation Disorder
MeSH Terms: conditions — Intestinal Pseudo-Obstruction; Nausea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Group that performed abdominal exercise for 1 week before operation.
  Interventions: Procedure: Abdominal Exercise (digital rectal stimulation, abdominal massage)
- Control Group (No Intervention): Group without preoperative abdominal exercise.

INTERVENTIONS:
Procedure: Abdominal Exercise (digital rectal stimulation, abdominal massage) — The recommended bowel exercise program consisted of three steps:
  1. Patients will perform a 2-3 minute massage starting from the cecum approximately 20-30 minutes after breakfast, moving along the colon.
  2. Patients will assume a suitable position and perform circular massage on the anal walls with their finger for approximately 30 seconds (digital rectal stimulation).
  3. Patients will try to defecate while sitting on the toilet.
  Arms: Exercise Group

SUMMARY:
Gastrointestinal dysfunction is a common complication after abdominal gynecologic oncology surgery. There are numerous studies in the literature addressing the management of bowel function in the postoperative period. Unfortunately, the strategies in the literature are not one hundred percent successful, and complete prevention of postoperative bowel dysfunction cannot be achieved. There is no study in the literature demonstrating that abdominal exercises given to patients undergoing surgery for gynecological malignancies in the preoperative period improve gastrointestinal function in the postoperative period.

The aim of this study is to evaluate the effect of an exercise plan, including abdominal massage and rectal digital stimulation, performed before gynecologic oncology surgery on postoperative bowel functions.

DETAILED DESCRIPTION:
This randomized study was approved by the Tepecik Training and Research Hospital Ethics Committee and conducted between January 1, 2023, and August 31, 2023. Patients diagnosed with gynecologic malignancies at our center were included in the study. Patients in the study group were provided with abdominal exercises one week before surgery, and they practiced exercises that included abdominal massage and rectal digital stimulation during the week leading up to the operation. Patients who did not perform exercises were included as the control group.

Participants were randomized after obtaining written informed consent forms. Patients with an operation plan were assigned to one of the two groups through randomization by the principal investigator. Group 1 patients constituted the control group, while Group 2 consisted of patients who regularly performed the recommended bowel exercise program every morning one week before the surgery. The recommended bowel exercise program was explained in detail to patients by the responsible researcher on the day of their preoperative anesthesia preparations (at least 10 days before the surgery) in the pre-op preparation room, accompanied by visual presentations. The recommended bowel exercise program consisted of three steps:

1. Patients will perform a 2-3 minute massage starting from the cecum approximately 20-30 minutes after breakfast, moving along the colon.
2. Patients will assume a suitable position and perform circular massage on the anal walls with their finger for approximately 30 seconds (digital rectal stimulation).
3. Patients will try to defecate while sitting on the toilet.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgery for endometrium, cervical and ovarian cancer indications,
* Patients with American Society of Anesthesiologists (ASA) score 1 or 2

Exclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) score 3 or 4
* Those with inflammatory bowel disease,
* Those who have abdominal fluid severe enough to prevent exercise,
* Patients with liver, kidney and thyroid function disorders,
* Patients with orthopedic problems affecting mobility,
* Patients with a history of abdominal bowel surgery,
* Those who received abdominal radiotherapy, hyperthermic intraperitoneal chemotherapy or neoadjuvant chemotherapy,
* Patients who had bowel injuries during surgery, bowel resection, anastomosis or colostomy,
* Patients who underwent Hipec,
* Patients who underwent relaparotomy before discharge due to reasons such as bleeding or evisceration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study was conducted in patients undergoing gynecologic oncology surgery.
Enrollment: 120 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
First exhaust and defecation time | postoperative period, an average of 15 days
  Postoperative time to first exhaust and defecation refers to the time elapsed from the end of the surgery to the first occurrence of gas and defecation.
Bowel Sounds | postoperative period, an average of 15 days
  Time to the return of bowel sounds is determined by researchers listening to bowel sounds with a stethoscope every 4 hours starting 8 hours after the surgery. It is based on the time when the first occurrence of 3-5 bowel sounds per minute is detected.
Solid food tolerance | postoperative period, an average of 15 days
  Duration of solid food tolerance is recorded as the time during which the patient can tolerate any food that requires chewing after surgery, without experiencing symptoms such as nausea or vomiting within 2 hours of consumption.
Length of hospital | postoperative period, an average of 15 days
  Duration of postoperative hospitalization.

SECONDARY OUTCOMES:
Postoperative gastrointestinal symptoms | postoperative period, an average of 15 days
  Abdominal pain, abdominal distension and nausea/vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffer Sancı, Study Director — Tepecik Training and Research Hospital
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No